CLINICAL TRIAL: NCT02668510
Title: A Randomized Controlled Pilot Trial Comparing Extracorporeal Shock Wave Therapy With Platelet Rich Plasma Versus Extracorporeal Shock Wave Therapy in a High Demand Cohort With Resistant Plantar Fasciitis
Brief Title: RCT Comparing ESWT With PRP for Plantar Fasciitis in High Demand Cohort
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Withdrawn as researcher left before data collection could be completed
Sponsor: Edna Rath (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Edna Rath, Human Protection Director, William Beaumont Army Medical Center
Organization: William Beaumont Army Medical Center (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 16/03
Record Dates: First submitted 2016-01-26; First posted 2016-01-29 (Estimated); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Fasciitis, Plantar
Keywords: Heel Pain; extracorporeal shock wave therapy; ESWT; shock wave; Soldiers; Platelet rich plasma; PRP; Autologous conditioned plasma; Military
MeSH Terms: conditions — Fasciitis, Plantar | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Platelet Rich Plasma Injection Group (Experimental): shockwave therapy within standard of care using Ossatron system with intervention injection of platelet rich plasma (PRP) using Arthex system, into the plantar fascia at the calcaneal origin
  Interventions: Biological: platelet rich plasma
- Placebo injection group (Placebo Comparator): shockwave therapy with placebo normal saline injection
  Interventions: Drug: Normal saline

INTERVENTIONS:
Biological: platelet rich plasma — immediately following shockwave therapy the injection of PRP derived from subjects own blood using Arthex double syringe system will be injected at the origin of the plantar fascia at the calcaneous
  Other Names: PRP
  Arms: Platelet Rich Plasma Injection Group
Drug: Normal saline — placebo injection of normal saline immediately following shockwave therapy
  Other Names: Placebo
  Arms: Placebo injection group

SUMMARY:
A Randomized Controlled Pilot Trial Comparing Extracorporeal Shock Wave Therapy with Platelet Rich Plasma versus Extracorporeal Shock Wave Therapy in a High Demand Cohort with Resistant Plantar Fasciitis

DETAILED DESCRIPTION:
The purpose of this proposal is to perform a high-quality pilot study testing the efficacy of ESWT in combination with PRP for the management of resistant plantar fasciitis. We endeavor to determine if the pilot evidence supports a large, randomized study; and to conduct a power analysis for the follow-on study. The proposed pilot study will be a prospective double-blinded randomized controlled trial comparing pain and functionality at the 3 week, 6 week, 12 week and 6 month marks between extracorporeal shock wave therapy (ESWT) with platelet rich plasma (PRP) injection versus extracorporeal shock wave therapy with placebo injection of normal saline.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Patients that are already selected for ESWT for the treatment of resistant plantar fasciitis as part of clinical care under the doctor-patient relationship
* X-ray imaging studies (Plain radiographs) documenting no additional sources for heel pain within 12 months(all x-rays were conducted as part of standard of care and no radiation will be specific to the research study)
* Active Duty Soldier as they are a high demand cohort with increased frequency of plantar fasciitis compared to the general population as outlined by Scher et al.
* Previously tried conservative management meeting referral to Orthopaedics: Pain medications, taping, orthoses, night splinting or physical therapy
* Body Mass Index (BMI) <40kg/m2

Exclusion Criteria:

* • History of trauma* or previous injury to heel requiring operative intervention

  * All Soldiers pending medical board evaluation or punitive action
  * History of connective tissue disorder (e.g., Marfan's Syndrome, Ehlers-Danlos disease, Rheumatoid Arthritis, etc.)
  * Leaving the geographical area permanently or for extended periods of time forcing loss to follow up
  * Treatment for plantar fasciitis with injection within the last 6 months
  * Surgical indication or internal derangement of the foot
  * Chronic pain conditions
  * Pregnancy
  * Tarsal tunnel syndrome
  * Baxter's neuritis
  * Rigid flat foot
  * Active infection of the Foot overlying the injection area
  * Use of immunomodulators, immunosuppressives, or chemotherapeutic agents
  * Allergy or hypersensitivity to any of the proposed treatment medications
  * Any other clinically significant acute or chronic medical conditions (e.g., bleeding disorder) that, in the judgment of the Investigator, would preclude the use of a PRP or that could compromise patient safety, limit the patient's ability to complete the study, and/or compromise the objectives of the study.

    * Trauma for this research study is defined as a specific event or mechanism of injury, such as a direct blow or twisting injury of the foot that initiated the onset of heel pain. The insidious onset of heel pain with prolonged running or other physical activity is not defined as a traumatic event.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2023-12-11 (Actual); Study Completion 2023-12-11 (Actual)

PRIMARY OUTCOMES:
Visual analog scale (VAS) | 3, 6, 12, 24 weeks
  Decreased first step pain over time with single treatment of ESWT & PRP as measured by the VAS

SECONDARY OUTCOMES:
Functional Ankle Ability Measure (FAAM) | 3, 6, 12, 24 weeks
  functionality scale
Functional Ankle Ability Measure extended sports scale | 3, 6, 12, 24 weeks
  sports subscale for sport related activity
return to activity | 3, 6, 12, 24 weeks
  achieving minimal clinical important difference (MCID) on FAAM sport scale
repeat treatment threshold | 3, 6, 12, 24 weeks
  Decreased need for repeat ESWT as proven by achieving MCID on FAAM

CONTACTS AND LOCATIONS:
Overall Officials: Timothy B Pekari, DSc, Principal Investigator — WBAMC; Amanda L Allen, MD, Principal Investigator — WBAMC; Lola Norton, Study Director — WBAMC; Desiree d diebold, md, Principal Investigator — wbamc
Locations (1):
- William Beaumont Army Medical Center, El Paso, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Ogden JA, Cross GL, Williams SS. Bilateral chronic proximal plantar fasciopathy: treatment with electrohydraulic orthotripsy. Foot Ankle Int. 2004 May;25(5):298-302. doi: 10.1177/107110070402500504. PMID 15134609
- [Background] Chew KT, Leong D, Lin CY, Lim KK, Tan B. Comparison of autologous conditioned plasma injection, extracorporeal shockwave therapy, and conventional treatment for plantar fasciitis: a randomized trial. PM R. 2013 Dec;5(12):1035-43. doi: 10.1016/j.pmrj.2013.08.590. Epub 2013 Aug 22. PMID 23973504
- [Background] Aqil A, Siddiqui MR, Solan M, Redfern DJ, Gulati V, Cobb JP. Extracorporeal shock wave therapy is effective in treating chronic plantar fasciitis: a meta-analysis of RCTs. Clin Orthop Relat Res. 2013 Nov;471(11):3645-52. doi: 10.1007/s11999-013-3132-2. Epub 2013 Jun 28. PMID 23813184
- [Background] Martin RL, Irrgang JJ, Burdett RG, Conti SF, Van Swearingen JM. Evidence of validity for the Foot and Ankle Ability Measure (FAAM). Foot Ankle Int. 2005 Nov;26(11):968-83. doi: 10.1177/107110070502601113. PMID 16309613
- [Background] Metzner G, Dohnalek C, Aigner E. High-energy Extracorporeal Shock-Wave Therapy (ESWT) for the treatment of chronic plantar fasciitis. Foot Ankle Int. 2010 Sep;31(9):790-6. doi: 10.3113/FAI.2010.0790. PMID 20880482
- [Background] Yin MC, Ye J, Yao M, Cui XJ, Xia Y, Shen QX, Tong ZY, Wu XQ, Ma JM, Mo W. Is extracorporeal shock wave therapy clinical efficacy for relief of chronic, recalcitrant plantar fasciitis? A systematic review and meta-analysis of randomized placebo or active-treatment controlled trials. Arch Phys Med Rehabil. 2014 Aug;95(8):1585-93. doi: 10.1016/j.apmr.2014.01.033. Epub 2014 Mar 21. PMID 24662810
- [Background] de Mos M, van der Windt AE, Jahr H, van Schie HT, Weinans H, Verhaar JA, van Osch GJ. Can platelet-rich plasma enhance tendon repair? A cell culture study. Am J Sports Med. 2008 Jun;36(6):1171-8. doi: 10.1177/0363546508314430. Epub 2008 Mar 7. PMID 18326832
- [Background] O'Malley MJ, Vosseller JT, Gu Y. Successful use of platelet-rich plasma for chronic plantar fasciitis. HSS J. 2013 Jul;9(2):129-33. doi: 10.1007/s11420-012-9321-9. Epub 2013 May 18. PMID 24426857
- [Background] Ang TW. The effectiveness of corticosteroid injection in the treatment of plantar fasciitis. Singapore Med J. 2015 Aug;56(8):423-32. doi: 10.11622/smedj.2015118. PMID 26311907
- [Background] Scher DL, Belmont PJ Jr, Bear R, Mountcastle SB, Orr JD, Owens BD. The incidence of plantar fasciitis in the United States military. J Bone Joint Surg Am. 2009 Dec;91(12):2867-72. doi: 10.2106/JBJS.I.00257. PMID 19952249